CLINICAL TRIAL: NCT01120847
Title: PTSD, Sleep Disordered Breathing And Genetics: Effects On Cognition
Brief Title: Post Traumatic Stress Disorder (PTSD), Sleep Disordered Breathing And Genetics: Effects On Cognition
Status: Completed | Type: Observational
Sponsor: Stanford University (Other)
Collaborators: US Department of Veterans Affairs (U.S. Federal Agency)
Responsible Party: Principal Investigator, Jerome A Yesavage,, Professor, Stanford University
Other Study IDs: SU-06302009-2920
Record Dates: First submitted 2010-05-07; First posted 2010-05-11 (Estimated); Last update posted 2020-02-28 (Actual); Status verified 2020-02

CONDITIONS: Stress Disorders, Post-Traumatic
MeSH Terms: conditions — Stress Disorders, Post-Traumatic

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — blood or saliva
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Veterans with PTSD: No intervention; this is an observational study.
- Control group w/out PTSD: No intervention; this is an observational study.

SUMMARY:
The current research program aims to study how sleep disordered breathing, age and genetics affect memory in older adult veterans with Posttraumatic Stress Disorder (PTSD).

The study will help researchers and clinicians better understand the relationship among PTSD, sleep disordered breathing, genetics and memory function.

DETAILED DESCRIPTION:
The research project will clarify how sleep disordered breathing and Apolipoprotein (APOE) status affect cognitive decline in a population already at risk for accelerated decline-veterans with PTSD.

To fill this knowledge gap properly, we will conduct a longitudinal study and data include analytic techniques designed specifically to identify moderators and mediators of clinical change.

ELIGIBILITY:
Inclusion Criteria:

1. Age 55 years or older, male or female veterans of any racial or ethnic group.
2. PTSD subjects will be positive for lifetime PTSD, related to any past lifetime traumatic experience and have a diagnosis of current, chronic PTSD by the Clinician Administered PTSD Scale (CAPS) criteria with current CAPS score > 40
3. Capable of giving informed consent for the study
4. Sufficient visual and auditory acuity for cognitive testing

Exclusion Criteria:

Psychiatric Exclusions:

1. Current or lifetime history of any psychiatric disorder with psychotic features
2. Current or lifetime bipolar disorder or delusional disorder
3. Prominent suicidal or homicidal ideation
4. Current exposure to trauma or recent exposure to trauma in the past 3 months.
5. Currently or have within the past six months met DSM-IV criteria for drug or alcohol abuse or dependence (except nicotine).
6. Presence of alcohol intoxication (by breathalyzer) or alcohol withdrawal (by exam) during testing
7. Diagnosis of probable or possible dementia
8. Mini-Mental State Exam (MMSE) < 23
9. History of seizure disorder.

Medical/Medication Exclusions:

1. Acute illness or unstable chronic illness (e.g., history of severe liver disease (cirrhosis, esophageal varices, ascites, portal hypertension, hepatic encephalopathy). Clinical or laboratory evidence of active hepatic disease will be recorded.
2. History of neurologic (e.g., multiple sclerosis, seizure disorder, stroke, history of transient ischemic attacks) or systemic illness affecting central nervous system (CNS) function (e.g. liver failure, kidney failure, congestive heart failure, systemic cancer)
3. Unstable or severe cardiovascular disease
4. Unstable gastrointestinal disorder
5. Uncontrolled hypertension
6. Head injury within one year
7. Loss of consciousness >24 hrs
8. Use of systemic steroid medication (with the exception of Estrogen replacement therapy which is permissible)
9. Illiterate or unable to read or write English or are judged by the investigator to be unable or unlikely to follow the study protocol
10. Toxicology evidence of illicit substance use.

Ages: 55 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: US war Veterans with PTSD and possible sleep problems
Sampling Method: Non-Probability Sample
Enrollment: 324 (Actual)
Dates: Start 2004-09 (Actual); Primary Completion 2017-03-10 (Actual); Study Completion 2017-03-10 (Actual)

PRIMARY OUTCOMES:
Change in Rey Auditory Verbal Learning Test-Measures auditory learning and memory | annually
  This scale measures auditory learning and memory. The raw score range is 0-15 and scaled score range is 0-19.For raw and scaled scores, higher values represent a better outcome. Subscales are not combined to compute a composite score.

SECONDARY OUTCOMES:
APOE status | sample taken at entry into study.
  APOE allele

CONTACTS AND LOCATIONS:
Overall Officials: Jerome A Yesavage, Principal Investigator — Stanford University
Locations (1):
- VA Palo Alto Health Care System, Palo Alto, California, United States